CLINICAL TRIAL: NCT01074554
Title: Phase I/II Study of the Effects of Antibiotics on Sarcoidosis Pathogenesis
Brief Title: Trial of Antimycobacterial Therapy in Sarcoidosis
Acronym: CLEAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Wonder Drake, Associate Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 091103
Record Dates: First submitted 2010-02-08; First posted 2010-02-24 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-09

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; mycobacteria; cutaneous lesions
MeSH Terms: conditions — Sarcoidosis; Mycobacterium Infections | interventions — Levofloxacin; Ethambutol; Azithromycin; Rifampin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic Regimen (Experimental): The Antibiotic Regimen consists of Levaquin 750 mg loading on day 1, then 500 mg po QD and Ethambutol 15-25 mg/kg for a maximum of 1200mg QD and Azithromycin 500mg on day 1, then 250 mg po QD and Rifampin 5-10 mg/kg for a maximum of 300mg po QD.
  All four drugs are given concomitantly.
  Interventions: Drug: Antibiotic Regimen
- Placebo Regimen (Placebo Comparator): The placebo regimen consists of Lactose tablets, one for each antibiotic with equivalent pills
  Interventions: Drug: Placebo Regimen

INTERVENTIONS:
Drug: Antibiotic Regimen — Levaquin 750 mg loading on day 1, then 500 mg po QD Ethambutol 15-25 mg/kg for a maximum of 1200mg QD Azithromycin 500mg on day 1, then 250 mg po QD Rifampin 5-10 mg/kg for a maximum of 300mg po QD All four drugs are given concomitanly
  Other Names: Levaquin=Levofloxacin; Ethambutol=Myambutol; Azithromycin=Zithromax; Rifampin=Rifadin
  Arms: Antibiotic Regimen
Drug: Placebo Regimen — lactose control tablets; one for each antibiotic with equivalent pills
  Other Names: Lactose control tablets
  Arms: Placebo Regimen

SUMMARY:
Growing research from independent laboratories provide an association between mycobacteria and sarcoidosis. More recent immunologic and molecular studies demonstrate immune responses to mycobacteria virulence factors. The purpose of this study is to assess if administration of anti-mycobacterial drug therapy will aid in resolution of cutaneous sarcoidosis lesions.

DETAILED DESCRIPTION:
Independent molecular and immunologic investigations strengthen the association between mycobacterial antigens and sarcoidosis pathogenesis. Molecular analysis of sarcoidosis granulomas reveals the presence of Mycobacterium tuberculosis complex (MTB) DNA and proteins that are significantly absent from granulomatous controls. Mycobacterial DNA has been detected in cutaneous sarcoidosis lesions, in addition to systemic immune responses against mycobacterial antigens. Due to the association between sarcoidosis and mycobacterial antigens, we postulated that broad spectrum antimycobacterial therapy could lead to restoration of T cell function and clinical improvement of chronic cutaneous sarcoidosis lesions. We investigated the safety and efficacy of Concomitant Levofloxacin, Ethambutol, Azithromycin, and Rifampin (CLEAR) therapy among chronic cutaneous sarcoidosis subjects, with change in lesion diameter from baseline to completion of 8 weeks of therapy as the primary endpoint; we assessed for decreases in granuloma burden, if granulomas were evident upon histologic examination. Change in modified Sarcoidosis Activity Severity Index (SASI) was the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoidosis as defined by the ATS/ERS/WASOG statement on sarcoidosis as defined by the clinical presentation consistent with sarcoidosis, biopsy finding granulomas, and no alternative for the cause of the granulomas, such as tuberculosis
2. Patients must have chronic cutaneous skin lesions with or without taking chronic therapy (corticosteroids, methotrexate (max 10mg/week), azathioprine, hydroxychloroquine, cyclophosphamide, minocycline, doxycycline and chloroquine), in which the dose has not been altered in the 2 months prior to starting the study.
3. Subject has a diagnosis of cutaneous sarcoidosis for greater than 6 months with a Sarcoidosis Activity and Severity Index assessment score of at least 4. Diagnosis can be made by either:

   * Skin lesions characteristic of sarcoidosis and a biopsy showing granulomas with no evidence of mycobacteria, fungus, or malignancy.
   * A biopsy that does not show granulomas, but the patient has characteristic skin lesions and history of clinical features suggesting sarcoidosis (previous biopsy revealing noncaseating granuloma, bilateral hilar adenopathy, erythema nodosum, uveitis, raised ACE level, BAL lymphocytosis (CD4:CD8>3.5), panda/lambda sign on gallium scan)
   * Accepted clinical variants include, but are not necessarily limited to the following:

     * lupus pernio
     * nodular
     * subcutaneous
     * annular
     * angiolupoid
     * plaque
     * papular
     * lichenoid
     * psoriasiform
   * For purposes of this study "moderate to severe cutaneous sarcoidosis" is defined as the presence of sarcoidal skin lesions with any of the following features:

     * At least 5 easily visible facial lesions, or
     * Disease which involves > 3% BSA, or
     * Disease which confers functional impairment (e.g. nasal or visual field obstruction), or
     * Disease which confers significant symptoms of itching and/or pain.
4. If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or is using one of the following methods of birth control for the duration of the study and 90 days after study completion:

   * condoms, sponge, foams, jellies, diaphragm, or intrauterine device
   * contraceptives (oral or parenteral) for three months prior to study drug administration
   * a vasectomized sole partner
   * Females of childbearing potential must have a negative serum pregnancy test at screening visit.

Exclusion Criteria:

1. No consent/inability to obtain consent.
2. Age less than 18 years of age.
3. Inability to obtain biopsy or draw blood.
4. CPK, ALT or AST >5 times upper limit of normal (ULN)
5. Pregnancy or breast feeding.
6. Current use of medications metabolized by rifampin (See Appendix).
7. Allergy to macrolides, quinolones or rifamycins.
8. Visual Impairment as defined by differentiating colors.
9. Family or personal history of long QT syndromes.
10. Patients receiving another interventional investigational drug within the 30 days prior to dosing
11. Use of any investigational medication within the past 28 days prior to study enrollment.
12. Subject has been hospitalized for infection or received IV antibiotics within the previous 2 months prior to baseline.
13. Subject has a history of tuberculosis at anytime or close contact with a person with active tuberculosis within the previous 6 months, or persistent or active infections requiring hospitalization or treatment with IV antibiotics, IV antiretrovirals, or IV antifungals within 30 days of baseline, OR oral antibiotics, antivirals, or antifungals for purpose of treating infection, within 14 days of baseline.
14. Evidence of other active skin diseases or skin infections during screening that may interfere with evaluation of sarcoidosis.
15. Subject has an active infection requiring systemic antibiotics at time of screening
16. Subject has a history of listeriosis, treated or untreated tuberculosis, exposure to individuals with tuberculosis.
17. Subject has a variant of sarcoidosis that is not amenable to study evaluation, in the absence of chronic indurated lesions, such as:

    * Acute, "benign" sarcoid associated with erythema nodosum
    * Acute iritis
    * Ichthyosiform sarcoidosis
    * Hypo- or hyperpigmented macular sarcoidosis
    * Ulcerative sarcoidosis
    * Erythroderma
    * Alopecia
18. Patients otherwise unsuitable for participation in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wonder P Drake, MD, Principal Investigator — Vanerbilt University School of Medicine
Locations (1):
- Vanderbilt University School of Medicine, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Drake WP, Oswald-Richter K, Richmond BW, Isom J, Burke VE, Algood H, Braun N, Taylor T, Pandit KV, Aboud C, Yu C, Kaminski N, Boyd AS, King LE. Oral antimycobacterial therapy in chronic cutaneous sarcoidosis: a randomized, single-masked, placebo-controlled study. JAMA Dermatol. 2013 Sep;149(9):1040-9. doi: 10.1001/jamadermatol.2013.4646. PMID 23863960

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient who was randomized to the CLEAR regimen did not have lesions compatible with sarcoidosis at baseline. This patient did not proceed with study participation and was removed from number of patients that started the study.
Groups:
- Antibiotics: This study will compare the effects of antibiotics or placebo on resolution of cutaneous sarcoidosis lesions.
- Lactose Tablets: Patients who are randomized to control arm will receive an equivalent number of lactose tablets.
Period: Overall Study
Arm/Group | Antibiotics | Lactose Tablets
Started | 14 | 15
Completed | 11 | 11
Not Completed | 3 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics | Lactose Tablets | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [41 to 60] | 53 [42 to 57] | 53 [42 to 58]
Gender [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Size at the Completion of Antibiotic Therapy, Measured on a Continuous Scale; Change Will be Determined by Change in Diameter of the Lesions
Time Frame: Baseline to 8 weeks
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Antibiotic Regimen | Placebo Regimen
Number analyzed (Participants) | 14 | 15
mm | -8.4 (14) | 0.07 (32.)

2. Primary Outcome: Granuloma Burden
Description: Number of patients with a decrease in Granuloma Burden (only in those patients having granulomas present at baseline biopsy)
Time Frame: Baseline to 8 weeks
Measure: Number; unit: participants
Arm/Group | Antibiotic Regimen | Placebo Regimen
Number analyzed (Participants) | 10 | 7
participants | 7 | 0

3. Secondary Outcome: Change in Modified Sarcoidosis Activity and Severity Index (SASI) at Completion of Therapy.
Description: Characterization of lesion severity was conducted using Modified Sarcoidosis Activity and Severity Index (SASI), measuring erythema, induration and desquamation. The modification was that the same scale was applied to any part of the body, instead of the face alone. The scale range is 0 (no problem) to 72 (very severe).
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antibiotic Regimen | Placebo Regimen
Number analyzed (Participants) | 14 | 15
units on a scale | -2.9 (2.5) | -0.6 (2.1)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Antibiotics | Lactose Tablets
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics (N=15) | Lactose Tablets (N=15)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
insomnia (General disorders) | 1 (1) | 0 (0)
pill burden (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No